CLINICAL TRIAL: NCT02762955
Title: International Multi-center Comparative Randomized Double-blind Clinical Trial of Efficacy and Safety of BCD-057 (Adalimumab Produced by BIOCAD, Russia) and Humira® (Adalimumab Produced by Vetter Pharma-Fertigung Gmbh & Co KG, Germany) in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Comparative Clinical Trial of Efficacy and Safety of BCD-057 and Humira® in Patients With Moderate to Severe Plaque Psoriasis
Acronym: CALYPSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-057-2
Record Dates: First submitted 2016-03-31; First posted 2016-05-05 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
Keywords: adalimumab; biosimilar; BCD-057; psoriasis; tumor necrosis factor; monoclonal antibody
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-057 group (Experimental): BCD-057 group includes patients with moderate to severe plaque psoriasis, who will receive BCD-057 subcutaneously at a dose 80 mg on week 0, then at a dose 40 mg on weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21 and 23. Patients will be invited for randomization at week 24 (in order to keep the double-blind design of the study), but it will have a formal character (assignment of a new randomization number and lot). From week 25 patients of this group will continue to receive BCD-057 at a dose 40 mg on weeks 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and 51.
  BCD-057 is adalimumab biosimilar, monoclonal antibody to tumor necrosis factor alfa.
  Interventions: Biological: BCD-057
- Humira® group (Active Comparator): Humira® group includes patients with moderate to severe plaque psoriasis, who will receive Humira® subcutaneously at a dose 80 mg on week 0, then at a dose 40 mg on weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23. At week 24 participants will re-randomized (1:1) to treatment with Humira® or will transitioned to BCD-057. Patients will receive BCD-057 or Humira® at a dose 40 mg on weeks 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and 51.
  BCD-057 is adalimumab biosimilar, monoclonal antibody to tumor necrosis factor alfa.
  Humira® is original drug of adalimumab, monoclonal antibody to tumor necrosis factor alfa.
  Interventions: Biological: Humira®

INTERVENTIONS:
Biological: BCD-057 — BCD-057 is biosimilar of adalimumab (produced by BIOCAD).
  Other Names: adalimumab
  Arms: BCD-057 group
Biological: Humira® — Humira is the original adalimumab (produced by F. Hoffman-La Roche)
  Other Names: adalimumab
  Arms: Humira® group

SUMMARY:
CALYPSO clinical study is a phase 3 study which is carried out to establish the efficacy, safety and pharmacokinetic equivalence of BCD-055 (adalimumab, manufactured by JSC BIOCAD, Russia) and Humira® when used in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
CALYPSO study is the next step of clinical evaluation of adalimumab biosimilar manufactured by joint-stock company (JSC) BIOCAD, Russia.The aim of this study is to establish that BCD-057 is equivalent to Humira® in terms of efficacy, safety and pharmacokinetics when used by the standard regimen in patients with plaque psoriasis.

The study will enroll 344 patients with moderate to severe plaque psoriasis, who will be randomized into 2 groups (1:1 ratio): patients from the first group will receive BCD-057 subcutaneously (SC) at a dose 80 mg on week 0, then at a dose 40 mg on weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21 and 23. Then participants of this group will be invited for randomization at week 25 (in order to keep the double-blind design of the study), but it will have a formal character (assignment of a new randomization number and lot). Patients will continue to receive 40 mg of BCD-057 on weeks 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and 51.

Patients from the second group will receive Humira® subcutaneously (SC) at a dose 80 mg on week 0, then at a dose 40 mg on weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21 and 23. At week 25 participants will re-randomized (1:1) to treatment with Humira® or will transitioned to BCD-057.They will receive Humira® or BCD-057 at a dose 40 mg on weeks 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and 51.

ELIGIBILITY:
Inclusion Criteria:

* Patient had written informed consent.
* Age between 18 and 75 years.
* Patient has moderate to severe plaque psoriasis with stable course of the disease for 6 months
* Patient has had at least 1 course of phototherapy or systemic treatment for psoriasis or are candidates for such treatment in opinion of Investigator.
* BSA affected by psoriasis ≥ 10%, PASI score ≥ 12, sPGA score ≥ 3.
* Patient has hemoglobin ≥ 10 g/dl, leucocytes count ≥ 3 000/mcl, thrombocytes count ≥ 100 000/mcl, neutrophil count ≥ 2 000/mcl, aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase exceed 2,5 or less times the upper limit of the normal range creatinine less than 176,8 µmol/l, no serologic or virologic markers of hepatitis B virus and hepatitis C virus, negative urine pregnancy test, no signs of tuberculosis (negative tuberculosis skin test or negative quantiferon test. Patients can be included in they have positive tuberculin test, have had Bacteria Calmette-Guerin (BCG) vaccination and have negative Diaskintest or negative quantiferon test. Patients can be included if they have positive tuberculin test, have not been vaccinated with BCG and also patients with positive or uncertain quantiferon test/Diaskintest if they have documented adequate prophylaxis of tuberculosis finished before first adalimumab injection AND have documented absence of contacts with patients who have active tuberculosis AND have no signs of tuberculosis on chest X-Ray that was performed during 3 months before randomization)
* Patients are able to perform all procedures planed by protocol.
* Patients are ready for contraception with reliable methods starting 2 weeks before entering the study, and up to 4 weeks after the last dose of study drug.

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
* Previous receipt of adalimumab, history of use of any other biological anti-tumor necrosis factor-alpha therapy. Prior use of two or more biologics for treatment of psoriasis.
* Previous receipt of monoclonal antibodies if they were cancelled less that in 12 weeks before screening
* Patient is taking corticosteroids for up to 4 weeks before signing informed consent and during screening, disease-modifying drugs including methotrexate, sulfasalazin and cyclosporin for up to 4 weeks before signing informed consent, leflunomide, cyclophosphamide for up to 6 months before signing informed consent, phototherapy including selective phototherapy and photochemotherapy for up to 4 weeks before signing informed consent, live or attenuated vaccines for up to 8 weeks before signing informed consent.
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid phototherapy.
* Subject has a planned surgical intervention during the study or had surgical intervention less than 30 days prior to study.
* Subject has an active infection or history of infections as follows: any active infection for which systemic anti-infectives were used within 28 days prior to signing informed consent; a serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to signing informed consent; recurrent or chronic infections or other active infection that, in the opinion of the Investigator, might cause this study to be detrimental to the subject.
* Subject has known history of human immunodeficiency virus or any other severe immunodeficiency.
* Hepatitis B surface antigen or Hepatitis B core antigen or Hepatitis C antibody positivity at screening.
* History of tuberculosis.
* Positive results of rapid plasma reagin-test for T.pallidum at screening.
* Active ongoing diseases other than psoriasis that might confound the evaluation of the benefit of treatment of adalimumab or can increase risk of adverse reactions: acute inflammatory diseases or exacerbation of chronic diseases otherwise than psoriasis; stable ischemic heart disease III-IV functional class, unstable angina or history of myocardial infarction less than 1 year before the signing of informed consent; moderate to severe heart failure (New York Heart Association [NYHA] class III/IV; severe resistant arterial hypertension, atopic bronchial asthma, history of angiooedema, moderate to severe respiratory insufficiency, chronic obstructive lung disease 3-4 grade, decompensated diabetes mellitus, systemic autoimmune diseases, active neurologic disorders or their symptoms, other underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy.
* Subject has history of malignancy within 5 years EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, OR in situ breast ductal carcinoma.
* Subject has a history of hypersensitivity to the active substance or to any of the excipients of adalimumab or BCD-057 or other monoclonal antibodies.
* Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study.
* Subject has any mental illness, including severe depressive disorders and / or suicidal thoughts in history, which, in the opinion of the investigator, may create excessive risk to the patient or to influence the patient's ability to follow the protocol.
* History of drug addiction, alcoholism.
* Simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation; previous participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Ratio of patients with PASI75 response after 16 weeks of therapy | 16 weeks of therapy
  Ratio of patients who developed a decrease in Psoriasis Area Severity Index score by 75% or more (PASI75) after 16 weeks of therapy with adalimumab vs. baseline.

SECONDARY OUTCOMES:
PASI Improvement (%) after 16, 24, 33 and 55 weeks of therapy with adalimumab. | 16, 24, 33 and 55 weeks of therapy
  Percent improvement in Psoriasis Area Severity Index (PASI) after 16, 24, 33 and 55 weeks of therapy with adalimumab.
Ratio of patients with PASI75 response after 24, 33, 55 weeks of therapy | 24, 33 and 55 weeks of therapy
  Ratio of patients who developed a decrease in Psoriasis Area Severity Index score by 75% or more (PASI75) after 33, 55 weeks of therapy with adalimumab vs. baseline.
Ratio of patients with PASI50 and PASI90 response after 16, 33, 55 weeks of therapy. | 16, 24, 33 and 55 weeks of therapy
  Ratio of patients who developed a decrease in Psoriasis Area Severity Index score by 50% or more (PASI50) and Psoriasis Area Severity Index score by 90% or more (PASI90) after 16, 24, 33, 55 weeks of therapy with adalimumab vs. baseline.
Ratio of patients with sPGA response after 16, 33, 55 weeks of therapy | 16, 24, 33 and 55 weeks of therapy
  Ratio of patients who have Physicians Global Assessment (sPGA) score 0 or 1 after 16, 33, 55 weeks of therapy with adalimumab.
BSA Improvement (%) after 16, 24, 33, 55 weeks of therapy | 16, 24, 33 and 55 weeks of therapy
  Percent of body surface area (BSA), affected by psoriasis (measured by physician during physical examination of patient), after 16, 33, 55 weeks of therapy with adalimumab vs. baseline.
Change in SF-36 | Week 0 to Week 16; Week 16 to Week 55
  Change in Short Form-36 questionnaire (SF-36) from Week 0 to Week 16 and from Week 16 to Week 55.
Change in DQLI | Week 0 to Week 16; Week 16 to Week 55
  Change in Dermatology Quality of Life Index questionnaire (DLQI) from Week 0 to Week 16 and from Week 16 to Week 55.
Adverse events (AE) severity and frequency related to adalimumab | 16 and 55 weeks of therapy
Overall adverse events (AE) and serious adverse events (SAE) frequency | 16 and 55 weeks of therapy
Frequency of early withdrawal due to AE/SAE | 16 and 55 weeks of therapy
Ratio of patients with binding and neutralizing antibodies to adalimumab | 55 weeks
AUC(0-tau) of adalimumab after multiple adalimumab injections | 55 weeks
  Area under the plasma concentration versus time curve (AUC) 0-tau of adalimumab after multiple adalimumab injections
Cav,ss of adalimumab after multiple adalimumab injections | 55 weeks
  Average blood concentration of adalimumab in steady state conditions (Cav,ss)
Т½ of adalimumab after multiple adalimumab injections | 55 weeks
  Half-life (Т½) of adalimumab after multiple adalimumab injections
Vd of adalimumab after multiple adalimumab injections | 55 weeks
  Volume of distribution (Vd) of adalimumab after multiple adalimumab injections
Cl of adalimumab after multiple adalimumab injections | 55 weeks
  Clearance (Cl) of adalimumab after multiple adalimumab injections

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (1):
- BIOCAD, Saint Petersburg, Strelna, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samtsov AV, Bakulev AL, Khairutdinov VR, Kokhan MM, Korotaeva TV, Minullin IK, Vylegzhanina OA, Dubenskiy VV, Khalilov BV, Khotko AA, Zykova OS, Chumachenko IV, Lukyanov AM, Artemeva AV, Pukhtinskaia PP. Long-term data on the proposed adalimumab biosimilar BCD-057 in patients with moderate to severe psoriasis: A randomized controlled trial. PLoS One. 2022 Feb 7;17(2):e0263214. doi: 10.1371/journal.pone.0263214. eCollection 2022. PMID 35130291